CLINICAL TRIAL: NCT04656769
Title: Impact of Analgesia on Cancer Recurrence and Mortality Within Five Years After Stage I Non-Small Cell Lung Cancer Resection
Brief Title: Analgesia aNd caNcer recUrrence Lung cAncer Resection
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Luca Brazzi, Principal investigator, University of Turin, Italy
Other Study IDs: ANNULAR
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Recurrence Tumor; Opioid Use, Unspecified; Analgesia; Thoracic Surgery
Keywords: Recurrence tumor; Opioid use; Analgesia; thoracic surgery
MeSH Terms: conditions — Recurrence; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PERI group
  Interventions: Procedure: Peridural analgesia
- EV group

INTERVENTIONS:
Procedure: Peridural analgesia — We attempted to evaluate the effectiveness of peridural analgesia through cancer survival and recurrence outcomes.
  Groups: PERI group

SUMMARY:
The choice of analgesia after cancer surgery may play a role in the onset of recurrence, particularly opioids seem to play a role in the immune system by promoting cancer cell proliferation and migration. Based on this consideration, our aim was to assess the impact of perioperative analgesia's choice on cancer recurrence after curative surgery for Stage I Non-Small Cell Lung Cancer. The investigators retrospectively reviewed the records of patients who underwent lung resection for Stage I NSCLC between January 2005 and December 2012. Patients received analgesia either by peridural (PERI group) or, in case of patient refusal or failure in catheter positioning, intravenous analgesia with opioids (EV group). Follow-up was concluded in August 2019. The five-year cumulative incidence of recurrence and the overall survival were evaluated and adjusted with a propensity score matching methodology.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yrs
* Patients who underwent lung resection for Stage I NSCLC between January 2005 and December 2012

Exclusion Criteria:

* Age<18aa
* Pregnancy
* Day hospital patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent lung resection for Stage I NSCLC between January 2005 and December 2012
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of recurrence and the overall survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Luca Brazzi, Professor, Study Chair — University of Torino; Giulio L Rosboch, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza; Ilaria De Domenici, MD, Study Director — University of Torino; Edoardo Ceraolo, MD, Principal Investigator — A.O.U. Città della Salute e della Scienza
Locations (1):
- AOU Città della Salute e della Scienza di Torino, Torino, Italy